CLINICAL TRIAL: NCT04409652
Title: Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine
Brief Title: Head Position on Preventing Emergence Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Associate professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AJIRB-MED-OBS-20-055
Record Dates: First submitted 2020-05-25; First posted 2020-06-01 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Gallbladder Diseases
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): The endotracheal extubation is performed in head on bed without pillow.
  Interventions: Procedure: Head on bed
- Head elevation group (Active Comparator): The endotracheal extubation is performed in head elevation on pillow (slight flextion of neck on chest) .
  Interventions: Procedure: Head on pillow

INTERVENTIONS:
Procedure: Head on bed — During emergence, head is kept on bed without pillow.
  Arms: Control group
Procedure: Head on pillow — During emergence, head is kept on pillow.
  Arms: Head elevation group

SUMMARY:
The purpose of this study is to investigate the effect of head position on prevent the emergence cough followed by endotracheal extubation.

DETAILED DESCRIPTION:
During endotrachl intubaion, the sniffing postion is most commonly recommended. However, the head position to reduce the emergence cough followed by endotracheal extubation was not confirmed yet. Considering the endotracheal tube vector, head elevation with pillow is thought to be acceptable more.

ELIGIBILITY:
Inclusion Criteria:

* Operation schedule of laparoscopic cholecystectomy
* Must be performed under general anesthesia

Exclusion Criteria:

* BMI > 30 kg/m2
* Respiratory infection
* Uncontrolled hypertension

Ages: 19 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The severity of cough | during extubation
  0: no cough, 1:single 2: more than one episode of non-sustained cough, 3: sustained and repetitive cough

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine, Suwon, South Korea